CLINICAL TRIAL: NCT03729037
Title: Comparative Evaluation of Video-based On-line Course vs. Serious Game for Training Medical Students in Cardiopulmonary Resuscitation: a Randomized Trial
Brief Title: Cardiopulmonary Resuscitation Self-training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1818537
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Cardiopulmonary Arrest With Successful Resuscitation
Keywords: Virtual learning; Educational technology; Medical education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious game (Experimental): Intervention: CPR self-training with serious game.
  Interventions: Other: CPR self-training
- Training video (Active Comparator): Intervention: CPR self-training with Keynote presentation with the addition of voice-over narration.
  Interventions: Other: CPR self-training

INTERVENTIONS:
Other: CPR self-training

SUMMARY:
Participants were 45 first-year medical students randomly assigned to cardiopulmonary resuscitation (CPR) self-training using either a video-based presentation or a serious game developed in a 3D learning environment for up to 20 min. Each participant was evaluated on a written, multiple-choice test (theoretical test) and then on a scenario of cardiac arrest (practical test) before and after exposure to the self-learning methods.

DETAILED DESCRIPTION:
A prospective, simulation-based, randomised controlled trial was conducted. Participants were randomised to the video group watched a video-recorded lecture on the management of adult cardiac arrest, while participants randomised to the game group played a serious game on the same topic.

The video was developed based on a previously recorded Keynote presentation (version 6.6.2, Apple Inc.) with the addition of voice-over narration of the events. The video was edited to contain the same information as provided in the serious game. The learning environment simulated an urban public space where the player should identify a victim of cardiac arrest and perform CPR manoeuvres. The game was designed to be a CPR self-learning tool for both health professionals and the lay public. The game involved only one rescuer without access to a portable defibrillator. During the game, the player should identify the victim, diagnose cardiac arrest correctly and initiate CPR as early as possible. The actions of the player were guided throughout the game by step-by-step instructions that should be followed to save the victim's life and to score on the game. Whenever the manoeuvres were not performed correctly, the victim died and the game automatically restarted from the beginning.

After exposure to the self-learning methods, participants were reassessed individually for their theoretical knowledge on a written, 10-question, multiple-choice test (theoretical post-test) and for their practical performance by three examiners, blinded to group assignment, who independently rated the participants' actions on a 10-min simulated scenario of cardiac arrest using a CPR training manikin (practical post-test).

Simulated scenario The same simulated scenario was used for pre-exposure and post-exposure practical evaluation. When the student entered the simulation room, a manikin was lying on the floor, simulating a person lying on the street, unconscious, not responding to stimulation and with no respiratory effort or pulse. The student was alone without access to medical equipment such as a defibrillator. Participants were expected to recognise the cardiac arrest, call the emergency services, and initiate chest compressions and ventilations as soon as possible for at least two cycles. A 10-min time limit was set for each simulation session.

ELIGIBILITY:
Inclusion Criteria:

* Being a medical student;
* Voluntary participation;
* No previous participation in CPR training.

Exclusion Criteria:

* Previous participation in CPR training.
* Refusal to participate.
* Not being enrolled in medical school.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
American Heart Association (AHA) Guidelines for CPR | 2 hours
  Mean performance score of students on each (theoretical and practical) test for each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: David P Sena, MD, PhD, Principal Investigator — Pontificia Universidade Catolica do Rio Grande do Sul (PUCRS)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhanji F, Donoghue AJ, Wolff MS, Flores GE, Halamek LP, Berman JM, Sinz EH, Cheng A. Part 14: Education: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S561-73. doi: 10.1161/CIR.0000000000000268. No abstract available. PMID 26473002
- [Background] Thorne CJ, Lockey AS, Bullock I, Hampshire S, Begum-Ali S, Perkins GD; Advanced Life Support Subcommittee of the Resuscitation Council (UK). E-learning in advanced life support--an evaluation by the Resuscitation Council (UK). Resuscitation. 2015 May;90:79-84. doi: 10.1016/j.resuscitation.2015.02.026. Epub 2015 Mar 9. PMID 25766092